CLINICAL TRIAL: NCT03399396
Title: Increasing HPV Vaccination in Community-Based Pediatric Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamela Hull (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Pamela Hull, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 171793; 1R01CA207401-01A1 (NIH)
Record Dates: First submitted 2017-12-20; First posted 2018-01-16 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: HPV Vaccines
MeSH Terms: interventions — Papillomavirus Vaccines

STUDY DESIGN:
Intervention Model Description: Using a two-group, cluster randomized control trial (RCT) design, with the clusters being pediatric practices, practices will be randomized to two study arms representing two delivery modalities of the intervention: In-Person Coaching Arm and Web-Based Coaching Arm.
  The intervention targets the providers and staff in the pediatric practices to make changes aimed to improve their quality of care, and the study participants are the providers and staff (not patients). Individual patients will not be recruited or enrolled in the study, since the intervention is focused on QI and all patient vaccination outcome data will be collected via aggregated reports from the EHR or other clinical data systems (no individual patient-level private health information (PHI)). The study practices include approximately 190 providers (physicians, nurse practitioners, physician assistants) and 275 other staff (nurses, clinical support staff, administrative staff).
Masking Description: Due to the nature of the intervention, it is not possible to blind the practices or study staff to study arm allocation. To minimize bias, allocation will be masked until after baseline data collection of outcome measures, when it is time for each practice to initiate the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-Based Coaching (Experimental): Web-based delivery of practice facilitation for HPV vaccine
  Interventions: Behavioral: Practice facilitation for HPV vaccine
- In-Person Coaching (Experimental): In-person delivery of practice facilitation for HPV vaccine
  Interventions: Behavioral: Practice facilitation for HPV vaccine

INTERVENTIONS:
Behavioral: Practice facilitation for HPV vaccine — The practice facilitation intervention provides coaching support to pediatric practices to guide them through quality improvement projects to increase HPV vaccination rates.

SUMMARY:
The central goal of this study is to identify the optimal approach to implementing an evidence-based practice facilitation (PF) intervention for the uptake and completion of HPV vaccine among adolescents receiving care in the community, guided by implementation science theory.

AIM 1: Determine the clinical effectiveness and cost-effectiveness of two modalities for delivering a multi-component PF intervention to increase HPV vaccination initiation and completion in community-based pediatric practices. The investigators will compare the traditional In-person Coaching PF modality to a lower-resource Web-Based Coaching PF modality. The primary patient outcome is HPV vaccination. The investigators will also examine and compare the sustainability of practice changes on vaccination rates and the effects over time for each intervention modality.

AIM 2. Understand mechanisms of why the PF intervention may work better for some pediatric practices than others for HPV vaccination. The investigators will examine theory-based determinants at the organizational, provider, and patient levels that may mediate (explain) or moderate (change) the effects of the PF intervention on vaccination outcomes.

DETAILED DESCRIPTION:
Background:

The human papillomavirus (HPV) vaccine offers the unprecedented opportunity to prevent nearly all cervical and anal cancers and a high proportion of vaginal, oropharyngeal, vulvar and penile cancers, where HPV is the etiologic agent. HPV vaccination is recommended for all children ages 11-12, with catch up for females to age 26 and males to age 21. However, despite clear and indisputable value in cancer prevention, uptake and completion of the HPV vaccine series has lagged far behind the goal of 80%. Provider recommendation is the strongest determinant of HPV vaccination, but slow translation of guidelines for preventive services, such as immunizations, into practice is a known challenge. Practice Facilitation (PF), also called quality improvement coaching, is a multicomponent quality improvement intervention approach that has well-established efficacy, in which external support and resources are provided to build the internal capacity of practices to improve quality of care and patient outcomes.

Objectives:

The central goal of the study is to identify the optimal approach to implementing an evidence-based intervention for the uptake and completion of HPV vaccine among adolescents receiving care in the community, guided by implementation science theory.

AIM 1: Determine the clinical effectiveness and cost-effectiveness of two modalities for delivering a multi-component PF intervention to increase HPV vaccination initiation and completion in community-based pediatric practices.

The investigators will compare the traditional In-person Coaching modality to a lower-resource Web-Based Coaching modality. The primary patient outcome is HPV vaccination. The investigators will also examine and compare the sustainability of practice changes on vaccination rates and the effects over time for each intervention modality.

H1: Both interventions will result in significant increases in HPV vaccination from baseline over time.

H2: Increases in the rate of HPV vaccination will be higher and sustained for a longer period of time in the In-person Coaching PF Arm as compared with the Web-Based Coaching Arm.

H3: The Web-Based Coaching Arm will be more cost-effective than the In-person Coaching Arm.

AIM 2. Understand mechanisms of why the PF intervention may work better for some pediatric practices than others for HPV vaccination.

The investigators will examine theory-based determinants at the organizational, provider, and patient levels that may mediate (explain) or moderate (change) the effects of the PF intervention on vaccination outcomes.

H4: Adoption of changes (process variables) and patient factors will mediate effects of the intervention on HPV vaccination outcomes.

H5: Organizational factors, provider attitudes, and intervention characteristics will moderate intervention effects on HPV vaccination outcomes.

Implications:

The findings will inform organizations about which PF modality to use among their constituent practices to improve HPV vaccination rates, with potential for future national dissemination.

ELIGIBILITY:
Inclusion Criteria:

* All providers and staff at each practice

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Age-appropriate completion rate (ages 13-17) | Annually, up to 3 years post baseline
  Percentage of active patients ages 13-17 who completed the HPV vaccine series before 13th birthday

SECONDARY OUTCOMES:
Age-appropriate initiation rate (ages 13-17) | Monthly, up to 36 months post baseline
  Percentage of active patients ages 13-17 who received at least one dose of HPV vaccine before 13th birthday
Age-appropriate completion rate (at age 13) | Monthly, up to 36 months post baseline
  Percentage of active patients who turned age 13 who completed the HPV vaccine series before 13th birthday
Age-appropriate initiation rate (at age 13) | Monthly, up to 36 months post baseline
  Percentage of active patients who turned age 13 who received at least one dose of HPV vaccine before 13th birthday
Overall completion rate (ages 13-17) | Monthly, up to 36 months post baseline
  Percentage of active patients ages 13-17 who completed the HPV vaccine series at any age
Overall initiation rate (ages 13-17) | Monthly, up to 36 months post baseline
  Percentage of active patients ages 13-17 who received at least one dose of HPV vaccine at any age
Dose received rate (well visits) | Monthly, up to 36 months post baseline
  Percentage of well visits in which a dose of HPV vaccine was administered (1st, 2nd, or 3rd dose), among all well visits for active vaccine-eligible patients ages 11-17
Dose received rate (all visits) | Monthly, up to 36 months post baseline
  Percentage of visits in which a dose of HPV vaccine was administered (1st, 2nd, or 3rd dose), among all visits for active vaccine-eligible patients ages 11-17
Age at vaccination | Monthly, up to 36 months post baseline
  Average age at receipt of first HPV vaccine dose, among active patients ages 13-17 who received 1st dose
Time to series completion | Monthly, up to 36 months post baseline
  Average number of months from 1st dose to last dose of HPV vaccine, among active patients ages 13-17 who completed the series

OTHER OUTCOMES:
Documented recommendation rate (well visits) | Monthly, up to 36 months post baseline
  Percentage of well visits with documentation of HPV vaccine either administered, deferred or refused, among all well visits for active vaccine-eligible patients ages 11-17
Documented recommendation rate (all visits) | Monthly, up to 36 months post baseline
  Percentage of visits with documentation of HPV vaccine either administered, deferred or refused, among all visits for active vaccine-eligible patients ages 11-17
Bundling adolescent vaccines rate | Monthly, up to 36 months post baseline
  Percentage of visits in which HPV, meningococcal, and Tdap vaccines were administered, among all visits for active patients ages 11-12 in which Tdap was administered and patient was eligible for both HPV and meningococcal vaccines
Missed opportunities rate | Monthly, up to 36 months post baseline
  Percentage of non-well visits in which HPV vaccine was not administered, among all visits for active vaccine-eligible patients ages 11-17

CONTACTS AND LOCATIONS:
Overall Officials: Pamela C Hull, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected from providers and staff (surveys and interviews) will be made available to other researchers upon request. All individual identifiers will be stripped to ensure confidentiality and privacy of study participants.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon request
Access Criteria: Qualified researcher with IRB approval

REFERENCES:
- [Derived] Chang RS, Shing JZ, Erves JC, Du L, Koyama T, Deppen S, Rentuza AB, McAfee C, Stroebel C, Cates J, Harnack L, Andrews D, Bramblett R, Hull PC. Measurement of provider fidelity to immunization guidelines: a mixed-methods study on the feasibility of documenting patient refusals of the human papillomavirus vaccine. BMC Med Inform Decis Mak. 2022 Dec 22;22(1):339. doi: 10.1186/s12911-022-02083-2. PMID 36550466